CLINICAL TRIAL: NCT03208270
Title: Pilot Study of Antithrombin Supplementation During Extracorporeal Membrane Oxigenation
Brief Title: Antithrombin Supplementation in ECMO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Collaborators: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Responsible Party: Principal Investigator, Mauro Panigada, MD, MD, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GATRA2016; 2016-004534-23 (EudraCT Number)
Record Dates: First submitted 2017-07-01; First posted 2017-07-05 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antithrombin supplementation (Experimental): Patients randomized to the study group will receive supplementation of antithrombin concentrate to maintain a functional antithrombin level between 80%-120%.
  Interventions: Drug: Antithrombin supplementation
- No Antithrombin supplementation (Active Comparator): Patients randomized to the control group will never receive supplementation of antithrombin unless "heparin resistance" occurs.
  Interventions: Drug: No antithrombin supplementation

INTERVENTIONS:
Drug: Antithrombin supplementation — antithrombin concentrate will be supplemented to maintain a functional antithrombin level between 80%-120%
  Other Names: Antithtrombin
  Arms: Antithrombin supplementation
Drug: No antithrombin supplementation — supplementation of antithrombin will not be provided unless "heparin resistance" occurs
  Other Names: No antithrombin
  Arms: No Antithrombin supplementation

SUMMARY:
Bleeding is the most feared complication during extracorporeal membrane oxygenation (ECMO) and is associated with high dosing of heparin. There is no consensus on antithrombin (AT) supplementation during ECMO. However, AT is needed by heparin to properly anticoagulate. We hypothesize that maintaining normal antithrombin levels during ECMO is associated with a less heparin dosing and more adequate level of anticoagulation.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) is a life support for patients with severe acute respiratory failure when conventional treatments failed but it is accompanied by a significant risk of bleeding. Heparin is required during ECMO to avoid circuit thrombosis and its anticoagulant effect is strictly dependent on antithrombin (AT). AT also plays a central role in mediating inflammation. Acquired AT deficiency is common in patients on ECMO, arguably due to long term anticoagulation in addition to sepsis itself. Guidelines suggest to supplement AT in ECMO only when its deficiency coexists with heparin resistance. Few studies evaluated the effect of AT supplementation during ECMO without a consensus on the appropriate level to be maintained. AT supplementation increase anti-Factor Xa (anti-Xa) levels without increasing heparin dosage. This may have a clinical impact because risk of bleeding during ECMO is associated with higher heparin dosage.

We hypothesize that maintaining normal antithrombin activity levels (80%-120%) during ECMO is associated with: I. less heparin dosage, II. a more adequate level of anticoagulation, III. less hemostasis related complications, and IV. a lower level of inflammation.

Adult patients on veno-venous ECMO for respiratory failure will be randomized to maintain AT between 80% and 100% (study group) or no supplementation unless heparin resistance occurs (control group). Sample size of at least 20 patients per group (n=40) is calculated upon the primary outcome measure of reduction of heparin use in the study group compared to the control group. AT and anti-Xa will be measured before ECMO and daily while on ECMO. Anticoagulation will be guaranteed with unfractionated heparin infusion with a target aPTT 1.5-2X normal. Study will end at ECMO removal.

Consistent literature suggests that current ECMO anticoagulation strategies are suboptimal probably due to improper antithrombin supplementation. A normal antithrombin level could guarantee an adequate anticoagulation regimen.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring veno-venous ECMO for severe respiratory failure.

Exclusion Criteria:

* patients with pre-existent heparin-induced thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Amount of heparin | through study completion, an average of 10 days
  Heparin dosage to maintain aPTT ratio between 1.5-2

SECONDARY OUTCOMES:
Bleeding | through study completion, an average of 10 days
  Bleeding complications
Adequacy of anticoagulation | through study completion, an average of 10 days
  Adequacy of anticoagulation, assessed through Anti-Xa levels
thrombosis | through study completion, an average of 10 days
  Patient's or circuit thrombosis
transfusions | through study completion, an average of 10 days
  Blood products transfusion requirements

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Panigada, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Panigada M, Spinelli E, De Falco S, Consonni D, Novembrino C, Boscolo Anzoletti M, Panarello G, Occhipinti G, Dos Santos CC, Pesenti A, Arcadipane A, Grasselli G. The relationship between antithrombin administration and inflammation during veno-venous ECMO. Sci Rep. 2022 Aug 22;12(1):14284. doi: 10.1038/s41598-022-17227-7. PMID 35995816
- [Derived] Panigada M, Spinelli E, Cucino A, Cipriani E, De Falco S, Panarello G, Occhipinti G, Arcadipane A, Sales G, Fanelli V, Brazzi L, Novembrino C, Consonni D, Pesenti A, Grasselli G. Antithrombin supplementation during extracorporeal membrane oxygenation: study protocol for a pilot randomized clinical trial. Trials. 2019 Jun 11;20(1):349. doi: 10.1186/s13063-019-3386-4. PMID 31186035